CLINICAL TRIAL: NCT01377350
Title: Non-invasive Heart Failure Monitoring Using Novel Acceleration Sensors System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Shmuel Rispler, Rambam Health Care Campus, P.O.B. 9602, Haifa 31096, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0550-10ctil; ministry of health Israel (Other: ministry of health Israel)
Record Dates: First submitted 2011-05-18; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-03

CONDITIONS: Heart Failure
Keywords: Heart failure; monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- "Pneumedicare"s monitoring system (Experimental): Single arm study - "Pneumedicare"s monitoring system is used for monitoring heart failure patients
  Interventions: Device: "Pneumedicare"s monitoring system.; Device: "Pneumedicare"s monitoring system

INTERVENTIONS:
Device: "Pneumedicare"s monitoring system. — 50 patients hospitalized due to the decompensated HF are considered for entry. 3 patches will be attached to the patients' thorax that include motion sensors. The system will be attached to the patients at the start of treatment. Patient's signals will be recorded during the entire treatment in the hospital, to the point that there is an improvement in their health condition.
  Other Names: "Pneumedicare"s monitoring system for heart failure patients
Device: "Pneumedicare"s monitoring system — Non invasive clinical follow-up of patients with HF deterioration and improvement, by a device-based algorithm. The system comprises of patches attached to the patients' thorax that include motion sensors (Accelerometers) that measure the chest wall dynamics and the mechanics of lung inflation and deflation.
  Other Names: "Pneumedicare"s monitoring system for heart failure patients

SUMMARY:
The purpose of this study is to explore the feasibility of monitoring hemodynamic changes, which result from heart failure exacerbations, by recording the respiratory effort, chest wall dynamics and quantifying the development of dyspnea by using miniature mechanical sensors that are attaches to the chest.

DETAILED DESCRIPTION:
Pulmonary veins congestion and fine changes in alveolar transudative effusion accumulation affect lung mechanics (compliance) and the respiratory effort. Moreover, the associated state of oxygen de-saturation is compensated by an increase in the respiratory effort. These changes in the respiratory effort are reflected in chest wall dynamics and may provide the earliest non-invasive sign for lung congestion and deterioration in the heart failure.

The research system comprises of patches attached to the patients' thorax that include motion sensors (Accelerometers) that measure the chest wall dynamics and the mechanics of lung inflation and deflation. The signals are acquired by a miniaturized device that amplifies and samples the signals, stores and analyzes the data and displays the trends on the screen.

ELIGIBILITY:
Inclusion Criteria:

* Acute decompensated HF
* Decompensated chronic HF in patients with NYHA class III-IV symptoms
* Age over 20 years
* Ejection fraction reduced below 35% OR doppler evidence of impaired left ventricular diastolic filling

Exclusion Criteria:

* Inability or unwillingness to follow the study protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
earliest non-invasive signs for lung congestion and deterioration in the heart failure | 18 months
  Exploring the feasibility of monitoring hemodynamic changes, which result from heart failure exacerbations, by recording the respiratory effort, chest wall dynamics and quantifying the development of dyspnea by using miniature mechanical sensors that are attaches to the chest.

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Rispler, MD PhD, Principal Investigator — Rambam Medical Center Haifa Israel
Locations (1):
- Rambam Health Care Campus, Haifa, Israel